CLINICAL TRIAL: NCT02411708
Title: A Phase 2 Study of the Safety and Effectiveness of SANGUINATE™ in the Treatment of Vaso-Occlusive Crises in the Ambulatory Setting: A Placebo-Controlled, Single-Dose, Single-Blind Study in Adults With Sickle Cell Disease
Brief Title: Study of SANGUINATE™ In the Treatment of Sickle Cell Disease Patients With Vaso-Occlusive Crisis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGSC-005
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — PEGylated carboxyhemoglobin bovine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SANGUINATE (Experimental): 320 mg/kg
  Interventions: Drug: SANGUINATE
- Placebo (Placebo Comparator): Normal saline IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SANGUINATE — Single two-hour infusion of SANGUINATE
  Other Names: pegylated carboxyhemoglobin bovine
  Arms: SANGUINATE
Drug: Placebo — Single two-hour infusion of placebo
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Safety and effect of SANGUINATE on Sickle Cell Disease patients experiencing a vaso-occlusive crisis

DETAILED DESCRIPTION:
Patients who are experiencing a vaso-occlusive crisis will report to the clinic for treatment and screening into the SGSC-005 study. Patients who meet all inclusion/exclusion criteria will be randomized to receive either SANGUINATE 320 mg/kg or placebo (saline) over a 2 hour infusion period. Assessments of vital signs, ECGs, safety labs, adverse events as well as patient and physician questionnaires will be completed up to 6 hours after the start of the infusion. Patients will then be assessed for discharge either to home or admitted to the hospital for further treatment depending on their disease severity. Follow-up phone calls will be completed 24 hours and 7 days after initiation of treatment . A follow-up visit will be completed in the clinic at 72 hours after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Sickle Cell Disease (all genotypes),
3. Diagnosis of a severe vaso-occlusive crisis (VOC), based on the clinical judgement of the Investigator,
4. Participant needs to be admitted to the ambulatory site for treatment of VOC requiring IV pain medication,
5. Able to provide written consent,
6. Able to receive IV infusion of study drug.

Exclusion Criteria:

1. In the judgment of the Investigator, the participant is not a good candidate for the study,
2. An acute severe complication of SCD beyond VOC,
3. Pregnant or actively trying to become pregnant, or breastfeeding,
4. Participant had > 6 urgent visits for SCD complications in the prior 3 months,
5. Fewer than 30 days since any prior treatment with IV pain medication for VOC,
6. Onset of current acute painful crisis > 3 days prior to dosing,
7. Evidence of moderate to severe renal insufficiency (CrCl < 50 mL/min) or chronic kidney disease, or of moderate to severe hepatic disease (LFTs > 2 x ULN) based on past medical history,
8. Concurrent or prior treatment within 90 days with an investigational medication,
9. Abnormal ECG due to cardiac ischemia and/or atrial fibrillation of acute onset, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Time to readiness for discharge from ambulatory site | 7 Days
  Defined as the time from the start of study drug infusion until the time of participant's response that their pain episode has improved enough for discharge; investigator's assessment of participant's readiness for discharge; and participant no longer requires IV opioid administration

SECONDARY OUTCOMES:
Safety of treatment | 1 Day
  as determined by changes in vital signs, EKG, biochemical, hematological, and urinalysis measures, and reported AEs
Extent of reduction in pain score during ambulatory visit as assessed by the participant on a 10-point pain scale | 1 Day
Total pain treatment received including the opioid dose (mg/kg) received during ambulatory visit | 1 Day
Global assessment of the participant's improvement by the Investigator or study staff (at the time of readiness for discharge from the ambulatory visit, and at the 72-hour follow-up visit) | 7 Days
Reduction in the rate of recurrent ambulatory visit(s) for the VOC within 7 days post discharge | 7 Days
Reduction in the rate of hospitalization(s) for VOC after treatment with SANGUINATE and within 7 days post-discharge | 7 Days

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - FSCDR, Hollywood, Florida
  - Florida Health Tampa General Hospital, Tampa, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins Univeristy School of Medicine, Baltimore, Maryland
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No